CLINICAL TRIAL: NCT00027118
Title: A Prospective (Cohort) Study to Identify Factors Affecting Morbidity Following the Diagnosis and Treatment of Patients With Breast Cancer: A Multi-Institutional Study Between the National Institutes of Health (NIH) Rehabilitation Medicine Department (RMD) and the Walter Reed National Military Medical Center (WRNMMC) Breast Care Center (BCC)
Brief Title: Morbidity After Diagnosis and Treatment of Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 020045; 02-CC-0045; NCT00513838 (obsolete NCT alias)
Record Dates: First submitted 2001-11-20; First posted 2001-11-21 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2016-08-17

CONDITIONS: Breast Cancer; Shoulder; Lymphedema; Fatigue
Keywords: Shoulder; Breast Cancer; Physical Therapy; Lymphedema; Quality of Life; Breast Cancer Surgery; Healthy Volunteer; HV; Normal Control
MeSH Terms: conditions — Breast Neoplasms; Lymphedema; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will examine the frequency and severity of problems in women with breast cancer for 2 years following initial medical treatment, including:

* Physical impairments, such as loss of strength or flexibility, increased weight and swelling.
* Symptom distress, such as pain, fatigue and weakness.
* Functional limitations and disabilities, such as loss of independence in activities of daily living (e.g., grooming, bathing, dressing, driving a car), work and social and recreational activities.

It will identify factors associated with these problems and try to determine their relationship to them.

Patients 18 years of age and older with stage I, II, III or IV breast cancer may be eligible for this study. Women who have a breast biopsy negative for cancer will also be enrolled as control subjects. Participants will be drawn from patients referred to the National Naval Medical Center for diagnosis and treatment during 2001-2003.

Participants will be evaluated over a 2-year period during an initial baseline visit (before medical treatment or biopsy) and follow-up visits at 1, 3, 6, 12, 18 and 24 months following procedures:

* Interview about past medical history and present illness, social and recreational activities, functional independence at work and during activities of daily living.
* Completion of questionnaires including health survey, upper limb disability questionnaire, and physical activity questionnaire. (Questionnaires are completed only at baseline and 12 and 24 months after medical treatment begins.) The questionnaires take about 30 to 40 minutes to complete.
* Upper body examination, including pain measurement using a 10-point scale, active and passive range of motion measures, manual muscle testing measures using a 10-point scale, timed upper limb lift test, and measures of upper limb volume and girth.

DETAILED DESCRIPTION:
Patients and healthy participants will undergo an interview at the beginning of the study and 1,3,6,9, 12, 18 and 24 months and answer questions about their medical history; family history; current problem and treatment; pain history; and social, physical and recreational activities. At the visit, they will also undergo an upper body physical exam by a physical therapist. Patients and the healthy participants will also fill out questionnaires about arm disability, quality of life, and physical activity at the beginning of the study and at 12, 18, and 24 months.

ELIGIBILITY:
* INCLUSION CRITERIA:

Population/Subjects: Individuals with breast cancer are identified among the patient population at National Naval Medical Center (NNMC). Patients referred to the NNMC Breast Care Center) NNMC-BCC for diagnosis and management (surgical treatment and radiation treatment or chemotherapy) of histologically established breast cancer (stage I, II, III, or IV) during 2001-2003, are eligible to participate in the study.

Healthy female individuals will be controls.

Subjects must be over 18 years of age and post-puberty as breast cancer does not occur prior to puberty; and been seen pre-surgical or medical intervention for baseline measurements and agree to participate in six follow-up visits of 30-45 minutes in duration during the next two-years.

EXCLUSION CRITERIA:

Subject chooses to not participate in the study.

Subjects are unable to complete the clinical examination tests.

Subjects are unable to complete the questionnaires/surveys.

Subjects are under age 18.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2001-11-16; Study Completion 2016-08-17

PRIMARY OUTCOMES:
Upper limb strength | 1,3,6,9, 12, 18 24 months
Upper limb range of motion | 1,3,6,9, 12, 18 24 months
Upper limb volume | 1,3,6,9, 12, 18 24 months
Arm disability questionnaire | 0, 12, 18, 24 months
Quality of life questionnaire | 0, 12, 18, 24 months
Physical activity questionnaire | 0, 12, 18, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Minal Jain, R.P.T., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Naval Medical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] King KB, Nail LM, Kreamer K, Strohl RA, Johnson JE. Patients' descriptions of the experience of receiving radiation therapy. Oncol Nurs Forum. 1985 Jul-Aug;12(4):55-61. No abstract available. PMID 3847996
- [Background] Meyerowitz BE, Watkins IK, Sparks FC. Quality of life for breast cancer patients receiving adjuvant chemotherapy. Am J Nurs. 1983 Feb;83(2):232-5. No abstract available. PMID 6549885
- [Background] Carter BJ. Women's experiences of lymphedema. Oncol Nurs Forum. 1997 Jun;24(5):875-82. PMID 9201739